CLINICAL TRIAL: NCT05806879
Title: The Impact of Using Maternity Napkins on the Incidence of Vaginal Infections in the Post-partum Period: A Randomized Controlled Trial
Brief Title: Impact of Maternity Napkins on the Incidence of Vaginal Infections in the Post-partum Period
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Farheen Yousuf, Assistant Professor, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6367
Record Dates: First submitted 2022-04-01; First posted 2023-04-10 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: Vaginal Infection
Keywords: Maternal Mortality; Maternal Morbidity; Sanitary Napkin; Maternity Napkin
MeSH Terms: conditions — Vaginitis; Maternal Death

STUDY DESIGN:
Intervention Model Description: Participants undergoing delivery at the maternal and child health centre will be randomized into an intervention and control group using a random number generator. The ratio of exposed to unexposed sample will be 1:1. The participants will be followed for 42 days via bi-weekly visits by research assistants.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Maternity Napkins (Experimental): The intervention group will receive maternity napkins to manage postpartum lochia with the following specifications:
  * Length is 230-240mm, to be able to provide adequate coverage.
  * Width is 150-155mm with wings.
  * Thickness is 3-5mm.
  * The maternity napkin is curved to prevent leakage on the sides, has wings for secure attachment to the underwear and able to absorb 30-40 ml per minute
  Interventions: Other: Maternity Napkin
- Continued Use of Current Methods (No Intervention): The control group will continue to use their current indigenous methods for managing postpartum lochia.

INTERVENTIONS:
Other: Maternity Napkin — Use of maternity napkin with the following specifications (followed for 4.5 months)
  * Length is 230-240mm, to be able to provide adequate coverage.
  * Width is 150-155mm with wings.
  * Thickness is 3-5mm.
  * The maternity napkin is curved to prevent leakage on the sides, has wings for secure attachment to the underwear and able to absorb 30-40 ml per minute.
  Arms: Maternity Napkins

SUMMARY:
This randomized controlled trial will compare the incidence of vaginal infections in the post-partum period in women using sanitary napkins, with women using their current methods of managing lochia. 350 women will be recruited from a health center present in Badin, Sindh, and will be randomized into an intervention or control group. The intervention group will receive maternity napkins while the control group will continue to use their current method of lochia management. Symptoms of vaginal infection and patient comfort with the method of lochia management will be assessed by a questionnaire administered by a research assistant via bi-weekly visits. A self -administered low vaginal swab will also be obtained at each visit.

DETAILED DESCRIPTION:
This is a randomized controlled trial using two parallel groups. District Thatta is a rural area that is situated two hours north of Karachi by drive. The Department of Community Health Sciences at the Aga Khan University (AKU), Karachi is working at District Thatta at established sites. In the proposed study, we will enroll 300 subjects in total randomized to either treatment or standard of care arm in a 1:1 ratio.

Thirty-six maternity napkins (two packets) will be provided to each participant at the time of recruitment and will be restocked at each follow-up visit. The control group will continue to use their current indigenous methods for managing postpartum lochia.

The research assistants will visit participants bi-weekly to administer questionnaires regarding symptoms of vaginal infection and comfort with use of method for management of lochia and restock the maternity napkins in the intervention group. Women who are unable to self-administer the questionnaire due to high illiteracy rates in the community, will be read out the form by the research assistant and their responses will be recorded. The research assistant will also provide the participant with equipment for a low vaginal swab at each bi-weekly visit with directions for administering. Once the participant has self-administered it, the research assistant will collect the swab and drop it at the clinical site. Alternatively, women will be invited to maternal and health center where the sample will be collected by a trained research assistant. If there is microorganism growth on a low vaginal swab, the participant will be informed and provided free treatment at the maternal and child health center. Any complications that arises during treatment including but not limited to sepsis and mortality will be documented. Any concomitant treatment that the participant wishes to receive will be recorded and there will be no restrictions placed on it.

The randomization method will use permuted blocks of variable size, randomly varying from 2 to 6 participants. Stratification factors in the randomization will be on the basis of type of delivery: vaginal delivery and Caesarian section (C-section) delivery since C-section delivery may be associated with a higher incidence of vaginal infection. The allocation will be secured in a plain white envelope. The nurse will provide maternity napkins to the participants in the intervention group and assign unique study identification (ID) numbers to each participant.

Participants will be randomized into an intervention and control group. Written and informed consent will be obtained from the participants prior to enrolment. The consent form has been translated to Sindhi for the purpose of this study. A research team member will be available close by to provide any clarification necessary. For participants who are unable to read, the consent from will be read out to them and their consent will be marked by a research team member. All information regarding the participants will be stored in a secured container and entered into an excel sheet which will be password protected with limited access to the research team only. The participant will be assigned a subject ID number to maintain the anonymity. In case a reproductive tract infection is detected, participants will be provided treatment free of cost by an available doctor at the maternal and child health center where the childbirth occurred according to culture and sensitivity. Serious adverse events are not expected because of the intervention. However, in case of a non-urgent adverse event, the participant will be provided a contact number at the time of recruitment which they can call to report the outcome and schedule an appointment at the maternal and child health center. In case of an emergency, the participant will be requested to visit the maternal and child health center and receive treatment. Treatment costs will be covered in both situations. For protocol deviation, a question has been included in the bi-weekly follow-up questionnaire where participants can report a deviation.

Single data entry with visual comparison will be performed to minimize error. Then, 10-15 forms will be randomly selected from the sample and the data on them will be compared to the data entered in the system. The information entered in the excel spreadsheet will be password protected. There will be limited access to the data by the research team only. The data will be de-identified once data collection is complete to maintain privacy of the participants. Case report forms (CRFs) and vaginal swab specimens will be transported from Thatta, Pakistan to the research laboratory at AKU in Karachi, Pakistan. These specimens will have their unique identifier, demonstrating the protocol name and number, patient ID number and date of sample collection. No personal information will be available on the vaginal specimen containers. The association between patient IDs and names will be stored in a database at the research office (data management unit) at the AKU. The primary investigator at AKU will have access to this secure database only. The research staff at AKU will only have access to de-identified CRFs and specimens.

Baseline demographics including name, age, height, weight, education, monthly income, and employment will be noted. Past medical history including comorbidities, parity, obstetric history, and previous postpartum complications will also be inquired. Finally, current medication and hygiene practices will also be noted. These variables will be recorded by the research team member during the examination. At the time of recruitment, details of the procedure will also be recorded using the hospital records including method used for cord clamping, antiseptic use etc.

All analysis will be conducted using SPSS software version 19. Baseline characteristics will be presented separately for both arms as frequency and percentage for categorical variables, mean and standard deviation for normal continuous variables and median and interquartile range for continuous variables with skewed distribution.

ELIGIBILITY:
Inclusion Criteria:

* Women above the age of 18 years who are undergoing delivery (spontaneous, induced, or assisted vaginal delivery and caesarean delivery) at the Maternal and Child Health Center
* Women between 1-3 days of the postpartum period
* Women who would not otherwise use sanitary napkins during the postpartum period

Exclusion Criteria:

* Women who currently already use sanitary napkins to manage lochia or who have undergone a caesarean (C-section) delivery will be excluded from this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Presence of Culture Positive Vaginal Infection | 4.5 months
  Participants will perform a self-taken low vaginal swab (LVS) every 2 weeks (bi-weekly) for confirmation of vaginal infection. Self-taken LVS are a viable alternative to clinician-taken high vaginal swab (HVS) with comparable sensitivity for detecting infection. Growth of micro-organisms including: Gardnerella vaginalis, Mycoplasma hominis, Prevotella species, Mobiluncus species, Trichomonas vaginalis, Candida albicans, Candida krusei, Candida glabrata will constitute positive culture growth.

SECONDARY OUTCOMES:
Symptoms of Vaginal Infection | 4.5 months
  Itching, perceived foul smelling vaginal discharge, fever, and lower abdominal pain will be inquired during the follow up visit every 2 weeks (bi-weekly) by the research assistant using an adapted questionnaire. The questionnaire will be validated in our study population before administration. The questionnaires have been developed in English and will be translated to Sindhi, the native language.
Patient Comfort based on Means of Lochia Management | 4.5 months
  Comfort of the patient will be inquired and recorded during the follow-up visit every 2 weeks (bi-weekly) using an adapted Likert scale, with 1 being not comfortable, and 5 being very comfortable. Comfort will be assessed based on three components including comfort, perception and behavior. The questionnaires have been developed in English and will be translated to Sindhi, the native language, and validated in the study population before administration to the control and intervention group.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ali TS, Fikree FF, Rahbar MH, Mahmud S. Frequency and determinants of vaginal infection in postpartum period: a cross-sectional survey from low socioeconomic settlements, Karachi, Pakistan. J Pak Med Assoc. 2006 Mar;56(3):99-103. PMID 16696506
- [Background] Ghani N, Rukanuddin RJ, Ali TS. Prevalence and factors associated with postpartum vaginal infection in the Khyber Agency federally administered tribal areas, Pakistan. J Pak Med Assoc. 2007 Jul;57(7):363-7. PMID 17867261
- [Background] Boushra M, Carlson K, Rahman O. Postpartum Infection. 2025 Jul 6. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK560804/ PMID 32809639
- [Background] Ali TS, Sami N, Khuwaja AK. Are unhygienic practices during the menstrual, partum and postpartum periods risk factors for secondary infertility? J Health Popul Nutr. 2007 Jun;25(2):189-94. PMID 17985820
- [Background] Chauhan G, Tadi P. Physiology, Postpartum Changes. 2022 Nov 14. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK555904/ PMID 32310364
- [Background] Sami N, Ali TS, Wasim S, Saleem S. Risk factors for secondary infertility among women in Karachi, Pakistan. PLoS One. 2012;7(4):e35828. doi: 10.1371/journal.pone.0035828. Epub 2012 Apr 27. PMID 22558233
- [Background] Shamshad, Shamsher S, Rauf B. Puerperal sepsis--still a major threat for parturient. J Ayub Med Coll Abbottabad. 2010 Jul-Sep;22(3):18-21. PMID 22338409
- [Background] Ely JW, Rijhsinghani A, Bowdler NC, Dawson JD. The association between manual removal of the placenta and postpartum endometritis following vaginal delivery. Obstet Gynecol. 1995 Dec;86(6):1002-6. doi: 10.1016/0029-7844(95)00327-n. PMID 7501321
- [Background] Fikree FF, Ali T, Durocher JM, Rahbar MH. Health service utilization for perceived postpartum morbidity among poor women living in Karachi. Soc Sci Med. 2004 Aug;59(4):681-94. doi: 10.1016/j.socscimed.2003.11.034. PMID 15177827
- [Background] Hainer BL, Gibson MV. Vaginitis. Am Fam Physician. 2011 Apr 1;83(7):807-15. PMID 21524046
- [Background] Barnes P, Vieira R, Harwood J, Chauhan M. Self-taken vaginal swabs versus clinician-taken for detection of candida and bacterial vaginosis: a case-control study in primary care. Br J Gen Pract. 2017 Dec;67(665):e824-e829. doi: 10.3399/bjgp17X693629. PMID 29158246
- See also: Adika YVO, Apiyanteide JFA, Ologidi PW, Ekpo KE. Perception and behaviour on use of sanitary pads during menstruation among adolescent school girls in Bayelsa State , Nigeria. Adv Appl Sci Res [Internet]. 2011;2(6):9-15. — https://www.primescholars.com/articles/perception-and-behaviour-on-use-of-sanitary-pads-during-menstruation-among-adolescent-school-girls-in-bayelsa-state-nigeria.pdf
- See also: Pakistan Maternal Mortality Survey 2019 — http://dhsprogram.com/pubs/pdf/PR128/PR128.pdf